CLINICAL TRIAL: NCT01152424
Title: Usefulness of Exhaled NO in the Differential Diagnosis Acute Eosinophilic Pneumonia and Community Acquired Pneumonia
Brief Title: Usefulness of Exhaled NO in the Differential Diagnosis Acute Eosinophilic Pneumonia and Bacterial Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sei Won Lee/ Assistant Professor, Seoul National University Bundang Hospital
Other Study IDs: FeNO in AEP
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Acute; Eosinophilic Pneumonia
Keywords: Acute eosinophilic pneumonia; Exhaled nitric oxide
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute eosinophilic pneumonia
- Community acquired pneumonia

SUMMARY:
Acute eosinophilic pneumonia (AEP) is diagnosed by cell count analysis of bronchoalveolar lavage fluid. However, the performance of bronchoscopy is not easy for patients with AEP, because they usually have hypoxia. Exhaled nitric oxide (FeNO) is usually elevated in the patients with eosinophilic inflammation such as asthma, but there is no previous studies FeNO in the patients with AEP. Investigators hypothesized that FeNO elevated significantly in patients with AEP, and FeNO can be used as non-invasive diagnostic method in patients who are clinically suspected with AEP, especially when the performance of bronchoscopy is difficult.

ELIGIBILITY:
Inclusion Criteria:

* All patients who visited the study hospital with bilateral pneumonic infiltration.

Exclusion Criteria:

* Patients who do not agree with our study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who visited the study hospital with bilateral pneumonic infiltration.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The difference of FeNO in AEP and Community Acquired Pneumonia | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Capital Hospital, Seongnam, Gyeongi, South Korea

REFERENCES:
- [Derived] Lee JE, Rhee CK, Lim JH, Lee SM, Shim YS, Lee CT, Won Lee S. Fraction of exhaled nitric oxide in patients with acute eosinophilic pneumonia. Chest. 2012 May;141(5):1267-1272. doi: 10.1378/chest.11-1303. Epub 2011 Oct 20. PMID 22016484